CLINICAL TRIAL: NCT04680936
Title: Is Low Dose Dextrose Prolotherapy as Effective as High Dose Dextrose Prolotherapy in the Treatment of Lateral Epicondylitis?- A Double Blind- Ultrasound Guided- Randomized Controlled Study
Brief Title: Low and High Dose Dextrose Prolotherapy in the Treatment of Lateral Epicondylitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, YILDIZ GONCA DOGRU, RESIDENT OF PHYSICAL MEDICINE AND REHABILITATION, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 14
Record Dates: First submitted 2020-12-13; First posted 2020-12-23 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Lateral Epicondylitis
Keywords: prolotherapy; dextrose prolotherapy; tennis elbow; chronic lateral epicondylitis; dextrose therapy
MeSH Terms: conditions — Tennis Elbow | interventions — Glucose; Water; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- low dose dextrose arm (5% dextrose) (Active Comparator): Prolotherapy injection will be made with 5% dextrose solution for 3 sessions with 3 weeks intervals. 1ml solution will be given with 27 Gauge 1/2 inch needles in the sessions. Before the treatment, the examination and questionnaire data of the patient will be recorded.
  Interventions: Drug: Dextrose 5% in water
- high dose dextrose arm (15% dextrose) (Active Comparator): Prolotherapy injection will be made with 15% dextrose solution for 3 sessions with 3 weeks intervals. 1ml solution will be given with 27 Gauge 1/2 inch needles in the sessions. Before the treatment, the examination and questionnaire data of the patient will be recorded.
  Interventions: Drug: Dextrose 15 % in Water
- Isotonic saline arm (0.9% NaCl) (Active Comparator): Prolotherapy injection will be made with isotonic saline for 3 sessions with 3 weeks intervals. 1ml solution will be given with 27 Gauge 1/2 inch needles in the sessions. Before the treatment, the examination and questionnaire data of the patient will be recorded.
  Interventions: Drug: Isotonic sodium chloride solution

INTERVENTIONS:
Drug: Dextrose 5% in water — low dose dextrose solution
  Other Names: 5% dextrose solution
  Arms: low dose dextrose arm (5% dextrose)
Drug: Dextrose 15 % in Water — high dose dextrose solution
  Other Names: 15%dextrose solution
  Arms: high dose dextrose arm (15% dextrose)
Drug: Isotonic sodium chloride solution — isotonic saline solution
  Other Names: 0.9% NaCl solution
  Arms: Isotonic saline arm (0.9% NaCl)

SUMMARY:
Lateral epicondylitis (tennis elbow) is an enthesopathy seen in 1-2% of the population aged 30-65 years, which can occur in the lateral epicondyle origo of the extensor carpi radialis brevis and longus muscles, after frequently repetitive activities and can lead to limitations in the daily life activities of the patients. The diagnosis is made by anamnesis and clinical examination, cases that last more than 3 months are defined as chronic lateral epicondylitis. Treatment options are analgesics, non-steroidal anti-inflammatory drugs, hand-wrist splints, eccentric strengthening exercises for forearm muscles and wrist dorsiflexors, injection therapies, physical therapy agents such as therapeutic ultrasound, ESWT(extracorporeal shockwave therapy), low-level laser therapy, and surgery. Prolotherapy is a treatment method that is performed with repetitive injections of a small amount of irritant or sclerosing solutions such as hypertonic dextrose, phenol-glycerin-glucose, or sodium morrhuate and aims to activate the healing process by increasing the blood flow around the damaged tendinopathy or enthesopathy area with the effect of these solutions. Hypertonic dextrose solutions in concentrations ranging from 12.5-20% are frequently used in prolotherapy. Prolotherapy can be done with ultrasound guidance or by determining anatomical landmarks. The injection is applied to the annular ligament, lateral epicondyle, and supracondylar area where the forearm extensor muscles adhere. Injection side effects and complications are pain, bruising, muscle spasm, nerve or vessel damage at the injection site. Based on previous studies, the low dose of dextrose solutions (1%, 5%, and 10%) may have a similar effect with fewer side effects than higher concentrations of dextrose solutions (15%, 20%, 25%) and the low dose may have fewer cell damage. Thus, it may be possible to apply an effective treatment method with fewer side effects in the treatment of lateral epicondylitis. Also, in this study, the effect of inflammation created by injection of saline in one group and the inflammatory, proliferative and angiogenic effects of dextrose injected in other groups at different concentrations on the treatment outcome will be compared.

DETAILED DESCRIPTION:
Lateral epicondylitis (tennis elbow) is an enthesopathy seen in 1-2% of the population aged 30-65 years, which can occur in the lateral epicondyle origo of the extensor carpi radialis brevis and longus muscles, after frequently repetitive activities and can lead to limitations in the daily life activities of the patients.

The diagnosis is made by anamnesis and clinical examination, cases that last more than 3 months are defined as chronic lateral epicondylitis.

Treatment options are analgesics, non-steroidal anti-inflammatory drugs, hand-wrist splints, eccentric strengthening exercises for forearm muscles and wrist dorsiflexors, injection therapies, physical therapy agents such as therapeutic ultrasound, ESWT(extracorporeal shockwave therapy), low-level laser therapy, and surgery.

Prolotherapy is a treatment method that is performed with repetitive injections of a small amount of irritant or sclerosing solutions such as hypertonic dextrose, phenol-glycerin-glucose, or sodium morrhuate and aims to activate the healing process by increasing the blood flow around the damaged tendinopathy or enthesopathy area with the effect of these solutions. Hypertonic dextrose solutions in concentrations ranging from 12.5-20% are frequently used in prolotherapy.

Dextrose is an ideal proliferant agent due to its ability to dissolve in water, exists in the blood chemically, and to led safely apply to more than one place. It is known that hypertonic dextrose solutions dehydrate the cells in the injection area, cause local tissue trauma, attracts granulocytes and macrophages to the damaged area, and triggers healing. Prolotherapy can be done with ultrasound guidance or by determining anatomical landmarks. The injection is applied to the annular ligament, lateral epicondyle, and supracondylar area where the forearm extensor muscles adhere. Injection side effects and complications are pain, bruising, muscle spasm, nerve or vessel damage at the injection site.

Based on previous studies, the low dose of dextrose solutions (1%, 5%, and 10%) may have a similar effect with fewer side effects than higher concentrations of dextrose solutions (15%, 20%, 25%) and the low dose may have fewer cell damage. Thus, it may be possible to apply an effective treatment method with fewer side effects in the treatment of lateral epicondylitis. Also, in this study, the effect of inflammation created by injection of saline in one group and the inflammatory, proliferative and angiogenic effects of dextrose injected in other groups at different concentrations on the treatment outcome will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Those who admit Kirsehir Ahi Evran University Hospital and is diagnosed with lateral epicondylitis,
* Participants with unilateral or bilateral lateral epicondylitis and pain and functional limitations due to this condition,
* who can read and write in Turkish,
* participant's admission participating in the study,
* participants who do not have exclusion criteria,

Exclusion Criteria:

* receiving any injection therapy to the elbow area in the last 3 months,
* participants with complaints less than 3 months(acute lateral epicondylitis)
* previously surgery on the elbow area,
* having a history of acute trauma or fracture in the elbow area,
* have local dermatological problems,
* have a local infection in the treatment area,
* those who are allergic to dextrose,
* with coagulation disorders or using anticoagulant drugs,
* with an autoimmune disease,
* with type 1 or type 2 diabetes mellitus,
* have unregulated hypertension,
* have immune dysfunction,
* with malignancy or diagnosed with a malignancy in the last 5 years,
* pregnancy or lactation,
* having cervical radiculopathy in the same extremity,
* with cognitive dysfunction,
* patients with paralysis in the same extremity,
* lack of cooperation due to cognitive impairment,
* participant's refusal to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of prolotherapy injection on hand grip strength. | Change of the hand grip strength at baseline, 3 weeks and after the injection treatment (12th week).
  Evaluation of the effect of prolotherapy injection on hand grip strength Hand grip strength will be measured with Hand-Dynamometer, before injection treatment (pre-intervention), at the 3rd week (2nd session of treatment) and after the injection treatment (12th week).
Evaluation of elbow pain that develops at rest and movement before, during and after injection treatment. | Change in elbow pain at baseline, 3 weeks and after the injection treatment (12th week).
  Elbow pain at rest and movement will be assessed by Visual Analogue Scale, before injection treatment (pre-intervention), at the 3rd week (2nd session of treatment) and after the injection treatment (12th week).
Evaluation of elbow pain threshold, before, during and after injection treatment. | Change in elbow pain threshold at baseline, 3 weeks and after the injection treatment (12th week).
  Elbow pain threshold will be assessed by Pain Algometer, before injection treatment (pre-intervention), at the 3rd week (2nd session of treatment) and after the injection treatment (12th week).
Assessment of the effect of elbow pain on daily life activities. | Change of the effect of elbow pain on daily life activities at baseline, 3 weeks and after the injection treatment (12th week).
  Daily life activities will be measured with Quick-DASH(Disabilities of Arm, Shoulder and Hand) Questionnaire, before injection treatment (pre-intervention), at the 3rd week (2nd session of treatment) and after the injection treatment (12th week).

SECONDARY OUTCOMES:
Evaluation of the clinical improvement. | week 3 and 12
  Clinical improvement of the patients will be evaluated subjectively with the Global Disease Assessment Questionnaire, before injection treatment (pre-intervention), at the 3rd week (2nd session of treatment) and after the injection treatment (12th week).
Evaluation of the injection side effects and complications. | 12 weeks
  Side effects and complications that may occur after injection treatments will be evaluated and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: FIGEN TUNCAY, PROF.,M.D., Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kirsehir Ahi Evran University Hospital, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hauser RA, Lackner JB, Steilen-Matias D, Harris DK. A Systematic Review of Dextrose Prolotherapy for Chronic Musculoskeletal Pain. Clin Med Insights Arthritis Musculoskelet Disord. 2016 Jul 7;9:139-59. doi: 10.4137/CMAMD.S39160. eCollection 2016. PMID 27429562
- [Background] Tsai SW, Hsu YJ, Lee MC, Huang HE, Huang CC, Tung YT. Effects of dextrose prolotherapy on contusion-induced muscle injuries in mice. Int J Med Sci. 2018 Jul 30;15(11):1251-1259. doi: 10.7150/ijms.24170. eCollection 2018. PMID 30123064
- [Background] Sims SE, Miller K, Elfar JC, Hammert WC. Non-surgical treatment of lateral epicondylitis: a systematic review of randomized controlled trials. Hand (N Y). 2014 Dec;9(4):419-46. doi: 10.1007/s11552-014-9642-x. PMID 25414603
- [Derived] Ciftci YGD, Tuncay F, Kocak FA, Okcu M. Is Low-Dose Dextrose Prolotherapy as Effective as High-Dose Dextrose Prolotherapy in the Treatment of Lateral Epicondylitis? A Double-Blind, Ultrasound Guided, Randomized Controlled Study. Arch Phys Med Rehabil. 2023 Feb;104(2):179-187. doi: 10.1016/j.apmr.2022.09.017. Epub 2022 Oct 13. PMID 36243123